CLINICAL TRIAL: NCT02621515
Title: An Open-label, Single-arm, Phase II, Multicenter Study to Evaluate the Efficacy of Nivolumab/Ipilimumab Combination Therapy in Metastatic Melanoma Patients With Symptomatic Brain Metastases.
Brief Title: Nivo/Ipi Combination Therapy in Symptomatic Brain Metastases
Acronym: CA209-322
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: In the Netherlands we wanted to add pilimumab to nivolumab. This resulted in a very long METC procedure which resulted in a to slow inclusion rate.
Sponsor: University Medical Center Groningen (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 201500776
Record Dates: First submitted 2015-09-09; First posted 2015-12-03 (Estimated); Last update posted 2024-05-06 (Actual); Status verified 2024-05

CONDITIONS: Melanoma; Brain Metastasis
Keywords: Nivolumab; Brain metastasis; Melanoma
MeSH Terms: conditions — Melanoma; Brain Neoplasms | interventions — Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Nivolumab (Experimental): All patients in this trial will receive treatment with nivolumab for 24 months. Treatment will be discontinued if confirmed disease progression has been demonstrated, if unacceptable toxicity or intercurrent illness prevents further treatment, and when informed consent is withdrawn. After discontinuation of treatment, follow-up will start. Duration of follow-up depends on survival of patients, with a maximum of 24 months. Therefore the end of this study is determined as 24 months after the last patient in this trial has started follow-up, has died, withdraws consent or is lost to follow-up for a different reason
  Interventions: Drug: Nivolumab

INTERVENTIONS:
Drug: Nivolumab — All patients in this phase 2 trial will receive treatment with nivolumab, a monoclonal antibody against the PD1-receptor on T cells. Dosing will be based on patients' weight (3 mg/kg). It will be administered in an intravenous infusion every 2 weeks and for a maximum of 2 years.
  Other Names: Opdivo

SUMMARY:
The effect of nivolumab on symptomatic brain metastases is currently unknown. This phase 2 clinical trial will be the first to evaluate this intracranial effect in humans, with the aim to give these patients the possibility to be treated with anti-PD-1. Besides the objective response rate, long term benefits in this patient category will be evaluated by measuring survival in terms of progression free survival and overall survival. Furthermore safety and tolerability of administration of this drug in patients with symptomatic brain metastases will be studied, as this is the first study for nivolumab in this specific patient category.

DETAILED DESCRIPTION:
This study is an open label, single arm, phase II clinical trial of prospectively collected data evaluating efficacy and safety of nivolumab in metastatic melanoma patients with symptomatic brain metastases. It will be conducted in several study centers in the Netherlands.

Patients with radiologic evidence of brain metastases and who are eligible for treatment with nivolumab will be screened for inclusion.

All patients in this trial will receive treatment with nivolumab for 24 months. Treatment will be discontinued if confirmed disease progression has been demonstrated, if unacceptable toxicity or intercurrent illness prevents further treatment, and when informed consent is withdrawn. After discontinuation of treatment, follow-up will start. Duration of follow-up depends on survival of patients, with a maximum of 24 months. Therefore the end of this study is determined as 24 months after the last patient in this trial has started follow-up, has died, withdraws consent or is lost to follow-up for a different reason.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must sign informed consent prior to inclusion in this trial.
2. Subjects must be ≥18 years of age and competent to give informed consent.
3. Histologically confirmed stage IV melanoma.
4. At least one radiologic new lesion in the brain by MRI, which should be measurable by RANO-BM criteria (longest diameter ≥ 10 mm and perpendicular diameter ≥ 5 mm). Lesions with prior local treatment (i.e., SRT or surgical resection) can be considered measurable if there has been demonstrated progression since the time of local treatment. Leptomeningeal involvement is allowed, but could not be used as target lesion.
5. BRAF status is determined. If positive, initial treatment for maximal 8 weeks with BRAF-inhibitors is allowed.
6. Subjects must be treatment-naive to nivolumab. (also as adjuvant treatment)
7. Eastern Cooperative Oncology Group (ECOG) Performance Status of 0-1.
8. Subjects must have adequate organ function as defined by the following laboratory values (determined within 28 days prior to randomization/registration):

   * White blood cells (WBC) ≥ 2000 /µL
   * Absolute neutrophil count (ANC) ≥ 1500 /µL
   * Platelets ≥ 100 x103 /µL
   * Hemoglobin ≥ 9 g/dL or ≥ 5.6 mmol/L
   * Serum creatinine ≤ 1.5 times upper limit of normal (ULN) or creatinine clearance > 40 ml/min (using the Cockcroft-Gault formula)
   * Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 3 times ULN
   * Bilirubin ≤ 1.5 times ULN (Except patient with Gilbert Syndrome, who can have total bilirubin ≤ 3.0 mg/dL)
   * LDH < 2 times ULN
9. Female subjects of childbearing potential should have a negative urine or serum pregnancy test within 24 hours prior to receiving the first administration of nivolumab. Women with non-childbearing potential may be included if they are either surgically sterile or have been postmenopausal for ≥ 1 year.
10. Women of child-bearing potential (WOCBP) and men who are sexually active with WOCBP must agree to use appropriate method(s) of contraception. (see section 5.2)

Exclusion Criteria:

1. Prior treatment with an anti-PD-1, anti-PD-L1, anti-PD-L2 antibody. (also as adjuvant treatment)
2. Subjects who have not recovered to Common Terminology Criteria for Adverse Events (CTCAE) v4.0 grade 1 or better from adverse events due to previous cancer therapy.
3. Evidence for an active, known or suspected autoimmune disease. Subjects are permitted to enroll if they have vitiligo, type I diabetes mellitus, residual hypothyroidism due to autoimmune condition only requiring hormone replacement, psoriasis not requiring systemic treatment, or conditions not expected to recur in the absence of an external trigger.
4. Treatment with corticosteroids in an increasing dosage in the 7 days prior to the first administration of nivolumab. (A stable or decreasing dosage of ≤ 4 mg dexamethasone or equivalent is allowed. In addition, inhaled or topical steroids and adrenal replacement doses are permitted in the absence of active autoimmune disease.)
5. Previous malignancies (except non-melanoma skin cancers, in situ bladder cancer, gastric or colon cancers, cervical cancers/dysplasia or breast carcinoma in situ) unless a complete remission was achieved at least 1 years prior to study entry and no additional therapy is required or anticipated to be required during the study period.
6. Previous severe hypersensitivity reaction to treatment with another monoclonal antibody, or known hypersensitivity to study drugs components.
7. A positive test for hepatitis B virus surface antigen (HBV sAg) or hepatitis C virus ribonucleic acid (HCV antibody) indicating acute or chronic infection.
8. Known history of testing positive for human immunodeficiency virus (HIV) or known acquired immunodeficiency syndrome (AIDS).
9. Any serious or uncontrolled medical disorder or active infection that, in the opinion of the investigator, may increase the risk associated with study participation, study drug administration, or would impair the ability of the patients to receive protocol therapy.
10. A known psychiatric or substance abuse disorder that could interfere with cancer therapy.
11. Women of childbearing potential with a positive serum or urine pregnancy test (minimum sensitivity 25 IU/L or equivalent units of HCG) within 24 hours prior to the start of nivolumab.
12. Breastfeeding women.
13. Inability to comply with other requirements of the protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2016-08 (Actual); Primary Completion 2018-05-30 (Actual); Study Completion 2018-05-30 (Actual)

PRIMARY OUTCOMES:
The best overall response rate (BORR) of brain metastases to nivolumab will be assessed on Magnetic Resonance Imaging (MRI) using the Response Assessment in Neuro-Oncology Brain Metastases (RANO-BM) criteria. | 2 years
  Per patient, the BORR of brain metastases to nivolumab will be assessed in terms of complete response, partial response, stable disease and progressive disease. An MRI of the brain will be used for radiologic response evaluation. Response evaluation will be performed according to the RANO-BM criteria.

SECONDARY OUTCOMES:
The difference in BORR will be assessed between previously treated and previously untreated brain metastases using the RANO-BM criteria. | 2 years
The difference in BORR will be assessed between intracranial metastases on and extra-cranial metastases within the same patient, using the RANO-BM criteria and the Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 criteria respectively. | 2 years
  Evaluation of intracranial metastases will be performed using MRI. Evaluation of extracranial metastases will be performed using CT.
Duration of response (DOR) | 4 years
  DOR is defined as the time between the date of first documented response (CR or PR) to the date of the first documented progression as determined by the RANO-BM criteria, or death due to any cause, whichever occurs first.
Time to development of new brain metastases in responding patients | 4 years
  For all responding patients, the time between response to study treatment, as assessed on MRI using the RANO-BM criteria, occurence of new brain metastases will be measured.
Progression free survival | 4 years
  Progression free survival is defined as the time from first administration of nivolumab to the date of the first documented progression, as determined by the RANO-BM criteria, or death due to any cause, whichever occurs first.
Overall survival | 4 years
  Overall survival is defined as the time between the date of first administration of nivolumab and the date of death.
The number of patients with treatment related adverse events as assessed by CTCAE v4.0. | 4 years

CONTACTS AND LOCATIONS:
Overall Officials: Geke AP Hospers, Md PhD, Principal Investigator — University Medical Center Groningen
Locations (4):
- Netherlands (4):
  - Dutch Cancer Institute/ A v. Leeuwenhoek Hospital, Amsterdam
  - VU Medical Center, Amsterdam
  - University Medical Center Groningen, Groningen
  - Erasmus Medical Center, Rotterdam